CLINICAL TRIAL: NCT02312388
Title: Comparison of the Central Venous Catheter Insertion Techniques: the Thin-wall Needle Versus the Catheter-over-the-needle Technique in Children
Brief Title: Comparison of the Central Venous Catheter Insertion Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-1303-113-478
Record Dates: First submitted 2014-11-27; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Child; Surgery
Keywords: central venous catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catheter-over-the-needle technique (Experimental): to use the 22G angiocatheter for central venous catheterization
  Interventions: Other: catheter-over-the-needle technique
- Thin-wall needle technique (Experimental): to use the sharp hollow 23G needle for central venous catheterization
  Interventions: Other: Thin-wall needle technique

INTERVENTIONS:
Other: catheter-over-the-needle technique — using a 22 G Angiocath Plus™ catheter
  Other Names: modified Seldinger technique
  Arms: Catheter-over-the-needle technique
Other: Thin-wall needle technique — using 18 - 21 G introducer needle
  Other Names: Seldinger technique
  Arms: Thin-wall needle technique

SUMMARY:
The purpose of this study is to compare the differences in central venous catheter insertion time, success rate, and complication between thin-wall needle technique and catheter-over-the-needle technique for central venous catheterization in children.

DETAILED DESCRIPTION:
Catheterization was performed using ultrasound with an "out-of-plane" approach by inserting the introducer needle (thin-wall needle technique) or Angiocath Plus™ catheter (catheter-over-the-needle technique) in 45 - 60° to the patient's skin while viewing the vein in a cross section.

ELIGIBILITY:
Inclusion Criteria:

* surgery under general anesthesia
* require central venous catheterization

Exclusion Criteria:

* hematoma in central vein
* central vein anomaly
* catheterization site infection

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Guide-wire insertion time | interval between skin penetration and removal of the needle or catheter after guide wire insertion, an expected average of 80 seconds

SECONDARY OUTCOMES:
Time to first puncture of central vein | interval between skin penetration of the needle or catheter and flashback of blood, an expected average of 25 seconds
Total time of central venous catheter insertion | interval between skin penetration of the needle or catheter and installation of the indwelling catheter, an expected average of 3 minutes
Number of central vein puncture trial | up to 5 times, an expected average observation time of 25 seconds
Number of guide-wire insertion trial | up to 5 times, an expected average observation time of 80 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD. PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea